CLINICAL TRIAL: NCT03269214
Title: Does Topical Phenytoin Enhance Healing Process in Bisphosphonate-related Osteonecrosis of the Mandible. A Uni-blind Clinical Trial Study
Brief Title: Use of Topical Phenytoin in Bisphosphonate-related Osteonecrosis of the Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, associate professor of oral and maxillofacial surgery, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1396D22
Record Dates: First submitted 2017-08-27; First posted 2017-08-31 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Osteonecrosis Due to Drugs, Jaw
Keywords: osteonecrosis; mandible
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Intervention Model Description: Patients who had bisphosphonate-related osteonecrosis of the jaw of the mandible randomly allocated in 2 groups. Group 1 underwent debridement of necrotic bone and the involved area closed primary and in group 2 ,patients received topical Phenytoin 5%+ Tetracycline
Who Masked: Participant, Investigator
Masking Description: Neither patients nor investigators were unaware about treatment and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients underwent debridement of necrotic bone and the involved area closed primary
- treatment group (Experimental): Patients received topical Phenytoin 5%+ Tetracycline after debridement before final closure.
  Interventions: Drug: Topical Phenytoin 5%

INTERVENTIONS:
Drug: Topical Phenytoin 5% — Patients received topical Phenytoin 5%+ Tetracycline after necrotic bone debridement .
  Arms: treatment group

SUMMARY:
Patients who had bisphosphonate-related osteonecrosis of the jaw in stage II were allocated in two groups randomly : In group1, 10 patients underwent debridement and primary closer of the area,in group 2 , patients received Phenytoin + tetracycline topically in the debridement area.Wound dehiscence , infection and pain were in 1,6 and 12 months after treatment.

DETAILED DESCRIPTION:
All patients undergo surgical necrotic bone debridement in combination with antibiotic therapy (clindamycin 300 mg q8h) for 4 weeks . Patients who had BRON of the mandible randomly allocated in 2 groups. Group 1 underwent debridement of necrotic bone and the involved area closed primary and in group 2 ,patients received topical Phenytoin 5%+ Tetracycline. Patients were evaluated after 1(time1) ,6(time2) and 12(time 3) months.

The size of bone lesion was measured by using come beam computer tomography (CBCT).

Wound dehiscence (Stage 0 :No dehiscence ,Stage 1: less than 10 mm dehiscence,stage 2 : more than 10 mm dehiscence) Infection: Pus, sinus tract (Yes/NO) Pain according to visual analog scale (VAS) 0-10.In the third follow up time ( 12 months) ,the number of patients who were a time span of 3 months without clinical symptoms were documented in each group.

ELIGIBILITY:
Inclusion Criteria:

* Criteria of bisphosphonate-related Osteonecrosis in stage II
* need debridement and surgical intervention

Exclusion Criteria:

* Malignancy in the area
* History of chemotherapy ,
* diabetic mellitus
* HIV
* odontogenic infection or undergo dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Soft tissue healing | After one month
  Appropriate soft tissue healing was defined when no dehiscence occurred
Soft tissue healing | Six months after treatment
  Appropriate soft tissue healing was defined when no dehiscence occurred
Soft tissue healing | 12 months after treatment
  Appropriate soft tissue healing was defined when no dehiscence occurred
Pain | one month after treatment
  Based on visual analogue scale 0-10
Pain | Six months after treatment
  Based on visual analogue scale 0-10

SECONDARY OUTCOMES:
Infection | One month after treatment
  Any sign of pus or fistula tract in treatment area
Infection | Six months after treatment
  Any sign of pus or fistula tract in treatment area
Infection | 12 months after treatment
  Any sign of pus or fistula tract in treatment area

IPD SHARING:
Plan to Share IPD: No
We realize final results without any information about individuals who attended in this study

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376